CLINICAL TRIAL: NCT05069103
Title: ImplementatioN of Remote Surgical wOund Assessment During the coviD-19 pandEmic
Acronym: INROADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Medical Research Council (Other Government); ISLACARE LTD (12108076) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AC21032
Record Dates: First submitted 2021-10-05; First posted 2021-10-06 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2023-12

CONDITIONS: Surgical Site Infection
Keywords: Telemedicine; Implementation
MeSH Terms: conditions — Surgical Wound Infection | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Similar to the original TWIST trial, patients will receive access to the online tool hosted on the ISLA platform until postoperative day 30 which is composed of two parts:
  1. A series of simple questions related to the detection of surgical wound infection (e.g. redness, swelling, fluid leakage, etc). These questions would be expected to be routinely asked during in-person assessment, and these questions have been previously developed and tested within the TWIST trial (the only change being the addition of questions specifically relating to the change in these symptoms).
  2. At least one image of their surgical wound(s).
  Patients will receive automated requests via notifications asking to complete the online tool over the 30-day period (every 3 days +/- 1 day), however they may also complete the online form whenever wished.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Similar to the original TWIST trial, patients will receive access to the online tool hosted on the ISLA platform until postoperative day 30 which is composed of two parts:
  1. A series of simple questions related to the detection of surgical wound infection (e.g. redness, swelling, fluid leakage, etc). These questions would be expected to be routinely asked during in-person assessment, and these questions have been previously developed and tested within the TWIST trial (the only change being the addition of questions specifically relating to the change in these symptoms).
  2. At least one image of their surgical wound(s).
  Patients will receive automated requests via notifications asking to complete the online tool over the 30-day period (every 3 days +/- 1 day), however they may also complete the online form whenever wished.
  Interventions: Device: Intervention

INTERVENTIONS:
Device: Intervention — Similar to the original TWIST trial , patients will receive access to the online tool hosted on the ISLA platform until postoperative day 30 which is composed of two parts:
  1. A series of simple questions related to the detection of surgical wound infection (e.g. redness, swelling, fluid leakage, etc). These questions would be expected to be routinely asked during in-person assessment, and these questions have been previously developed and tested within the TWIST trial (the only change being the addition of questions specifically relating to the change in these symptoms).
  2. At least one image of their surgical wound(s).

SUMMARY:
This is a implementation research study of a surgical wound tele-monitoring online tool developed at the University of Edinburgh and demonstrated in the "Tracking wound infection with smartphone technology" (TWIST) randomised control trial (NCT02704897) conducted in NHS Lothian. The study design is based on the Medical Research Council (MRC) "Guidance for developing and evaluating complex interventions".

DETAILED DESCRIPTION:
Surgical site infection (SSI) is one of the most common complications following surgery with significant costs to patients and health systems. Earlier diagnosis and treatment of SSI can reduce its impact. The investigators have previously developed a unique remote wound surveillance tool in a University of Edinburgh research setting. The investigators have demonstrated in a previous randomised controlled trial (NCT02704897), that wound infection can be diagnosed sooner (in the first 7 days postoperatively) when this tool is used.

This 12-month implementation research study will be conducted across the general surgical departments of the Royal Infirmary of Edinburgh and the Western General Hospital (two large tertiary hospitals). Informed consent will be required from all patients prior to enrolment, with a target of 200 patients recruited.

All data during the study will be collected via online forms hosted on the ISLA care platform, self-submitted by patients based on their own concerns with their wound or prompted by a routine request to complete. These forms are based on the smartphone-delivered wound assessment model developed and delivered in the TWIST trial (based on the Center for Disease Control and Prevention (CDC) classification criteria, and the ASEPSIS model (Additional treatment, Serous discharge, Erythema, Purulent exudate, and Separation of the deep tissues, the Isolation of bacteria, and the duration of Inpatient Stay)). Participants will be asked to upload at least one photograph of their wound each time they use the smartphone-delivered wound assessment tool. Participants will be sent one (1) reminder notification the following day if they have not completed a requested response.

On postoperative day 30-day, patients will be requested to complete an online questionnaire based on two validated questionnaires: Bluebelle Wound Healing Questionnaire (WHQ) and Telehealth Usability Questionnaire. Furthermore, a subset of patients will be asked to indicate their interest to take part in a separate semi-structured interview regarding their experience within the study, and views of telemedicine in routine postoperative care (target 20 patients).

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 16 years) with the capacity to provide informed consent
* Patient undergoing abdominal surgery who own a smartphone capable of accessing and completing the online response form

Exclusion Criteria:

* Any participants with self-reported impairment that would prevent use of the online questionnaires (and no alternative means for completion e.g. assistance from family or carers).

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Technology acceptance | 30 days
  Technology Intervention acceptance as measured by Telehealth Usability Questionnaire (TUQ)

SECONDARY OUTCOMES:
Health service usage | 30 days
  Attendance at community (general practice) or emergency hospital services (emergency department or the surgical treatment centre)
Time-to-diagnosis (days) of surgical-site infection | 30 days
  Time-to-diagnosis (days) of surgical-site infection (CDC criteria)
surgical-site infection interventions | 30 days
  Therapeutic intervention received for surgical site infection

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Western General Hospital, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
Anonomysed IPD shared for research purposes
Supporting Information: Study Protocol, Analytic Code
Time Frame: One year following publication
Access Criteria: Request from chief investigator (Professor Ewen Harrison)

REFERENCES:
- [Derived] McLean KA, Sgro A, Brown LR, Buijs LF, Mozolowski K, Daines L, Cresswell K, Potter MA, Bouamrane MM, Harrison EM. Implementation of digital remote postoperative monitoring in routine practice: a qualitative study of barriers and facilitators. BMC Med Inform Decis Mak. 2024 Oct 21;24(1):307. doi: 10.1186/s12911-024-02670-5. PMID 39434121
- [Derived] McLean KA, Sgro A, Brown LR, Buijs LF, Daines L, Potter MA, Bouamrane MM, Harrison EM. Evaluation of remote digital postoperative wound monitoring in routine surgical practice. NPJ Digit Med. 2023 May 5;6(1):85. doi: 10.1038/s41746-023-00824-9. PMID 37147462